CLINICAL TRIAL: NCT02077608
Title: Effect of Hyaluronan Enriched Embryo Transfer Media on IVF Outcome
Brief Title: Hyaluronan in Embryo Transfer Media
Status: Completed | Type: Observational
Sponsor: Peter Fancsovits, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Peter Fancsovits, Ph.D., Senior Clincial Embryologist, Semmelweis University
Organization: Semmelweis University (Other)
Other Study IDs: SemmelweisU-002
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Infertility
Keywords: In vitro fertilization; Embryotransfer; Hyaluronan; Pregnancy rate; Implantation rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hyaluronan enriched transfer media: Embryos are incubated at least 10 minutes in hyaluronan enriched embryo transfer media before transfer
- Control group: Embryos are incubated in embryo transfer media containing low concentration of hyaluronan for at least 10 minutes before transfer

SUMMARY:
Prospective randomized double blind comparison of hyaluronan enriched embryotransfer media and conventional embryotransfer media in human IVF treatments. Embryos selected for transfer are incubated in a culture media containing high concentration of hyaluronan or low concentration of hyaluronan.

Primary outcome: implantation and pregnancy rates

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients
* entering in vitro fertilization treatment
* at least 1 embryo transferred

Exclusion Criteria:

* IVF treatment with donated oocytes
* No embryo available for transfer

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients entering in vitro fertilization and embryo transfer treatment
Sampling Method: Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2010-01; Primary Completion 2012-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 5 weeks after embryo transfer
  Number of clinical pregnancies (gestational sacs visible by ultrasound examination) divided by the number of embryotransfers
Implantation rate | 5 weeks after embryotransfer
  Number of embryos implanted (No. of gestational sacs) divided by the number of embryos implanted

SECONDARY OUTCOMES:
Multiple pregnancy rate | 5 weeks after embryotransfer
  Number of multiple pregnancies divided by the number of embryotransfers
Delivery rate | 40 weeks after embryo transfer
  Number of delivery divided by the number of embryo transfers

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fancsovits, Ph.D., Study Chair — Semmelweis University First Department of Obstetrics and Gynecology; Janos Urbancsek, MD, Ph.D., Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology; Adam Lehner, MSc, Principal Investigator — Semmelweis University First Department of Obstetrics and Gynecology
Locations (1):
- Semmelweis University First Department of Obstetrics and Gynecology, Budapest, Hungary

REFERENCES:
- [Result] Bontekoe S, Heineman MJ, Johnson N, Blake D. Adherence compounds in embryo transfer media for assisted reproductive technologies. Cochrane Database Syst Rev. 2014 Feb 25;2014(2):CD007421. doi: 10.1002/14651858.CD007421.pub3. PMID 24567053